CLINICAL TRIAL: NCT03320785
Title: Circulating Markers in Preterm Infants With Perinatal and Neonatal Inflammation: An Observational Study
Brief Title: Circulating Markers in Preterm Infants With Perinatal and Neonatal Inflammation
Acronym: NEOINFLAM
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator unable to incorporate study and recruitments into clinical routines
Sponsor: Per Torp Sangild (Other)
Collaborators: Baoan Maternal And Child Health Care Hospital, Shenzhen, China (Unknown)
Responsible Party: Sponsor-Investigator, Per Torp Sangild, Professor, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: NEOINFLAM 2017
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Necrotizing Enterocolitis; Chorioamnionitis; Feeding Intolerance
Keywords: preterm infants; sepsis; chorioamnionitis; circulating markers
MeSH Terms: conditions — Sepsis; Enterocolitis, Necrotizing; Chorioamnionitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen whole blood and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Circulating markers to diagnose complications (sepsis, necrotizing enterocolitis) in preterm infants are often inaccurate, partly due to the lack of comprehensive studies with temporal evaluation from birth until a disease onset. The investigators plan to collect weekly blood samples of preterm infants from birth until 4 weeks of age to comprehensively characterize differential protein and epigenetic markers in infants with and without complications (sepsis, necrotizing enterocolitis, chorioamnionitis).

DETAILED DESCRIPTION:
Preterm infants (10% incidence worldwide), especially those who do not receive sufficient mother's own milk, are susceptible to infectious diseases including sepsis and necrotizing enterocolitis. Infants with history of prenatal inflammation including chorioamnionitis may be at higher risks of acquiring these infectious diseases. Limited knowledge is available regarding a comprehensive temporal profile of circulating markers in preterm infants from birth to disease onset. This current study aims to provide a comprehensive temporal profile of circulating markers, via -omic techniques (proteomics and/or epigenetics), during the first 4 weeks of life in preterm infants with various systemic complications. Thus, this will elucidate a profile of early markers consistently associated with pathological conditions in the whole study period. Depending on the outcome, a subsequent study for validation may be performed.

Primary objective: To characterize circulating markers associated with the early life complications including chorioamnionitis, LOS and NEC in preterm infants during the first four weeks of life.

Secondary objective: To characterize how different feeding regimes and diets may affect these markers during the first four weeks of life in preterm infants

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born before the complete 32 weeks of gestation
* Signed parental consent

Exclusion Criteria:

* Major congenital anomalies or birth defects

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study recruits very preterm infants (< 32 weeks of gestation) at the Department of Neonatology, Bao'An maternal and Child Health Hospital right after birth after screening inclusion and exclusion criteria. Information about maternal conditions (premature rupture of membranes or chorioamnionitis) and birth are collected but are not determining factor to recruit.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Circulating markers | From birth until 4 weeks of age or until discharge, whichever comes first
  Temporal profile of circulating markers are characterized from weekly collected blood samples (from birth until 4 weeks of age or until discharge, whichever comes first). Profiles are compared between:
  1. Infants without and with sepsis/NEC.
  2. Infants without and with clinical/histological chorioamnionitis.
  3. Infants receiving different type or amount of milk diets (e.g. mother´s own milk, donor milk, formula, fortifier)

CONTACTS AND LOCATIONS:
Overall Officials: Per T Sangild, PhD, Study Director — Rigshospitalet, Denmark
Locations (1):
- Shenzheng Baoan Maternity and Child Healthcare Hospital (SBMCH), Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The current clinical trial is a part of the NEOMUNE project. — http://neomune.ku.dk/

DOCUMENTS (1):
  • Study Protocol (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT03320785/Prot_000.pdf